CLINICAL TRIAL: NCT02255630
Title: The Effects of High-dose Salbutamol on Anaerobic Cycling Power
Brief Title: Anaerobic Power and Salbutamol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Natural Sciences and Engineering Research Council, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: H14-02788
Record Dates: First submitted 2014-09-16; First posted 2014-10-02 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Ergogenic Athletic Performance
Keywords: salbutamol; exercise-induced bronchoconstriction; anaerobic power

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Salbutamol inhalation (Experimental): Study participants will be exposed to 1600ug salbutamol 30min prior to exercise
  Interventions: Other: Cycling Exercise
- Placebo inhalation (Experimental): Study participants will be exposed to 1600ug salbutamol 30min prior to exercise
  Interventions: Other: Cycling Exercise

INTERVENTIONS:
Other: Cycling Exercise

SUMMARY:
Athletes using inhaled β2-adrenoreceptor agonists (IBAs) win a disproportionate number of medals. However, most previous research has shown that β2 agonists do not improve exercise performance in either asthmatic or non-asthmatic athletes. Although the majority of these studies do not show an ergogenic effect, the small number of studies with extended exercise bouts (~60 minutes) do show an advantage. The investigators believe that a controlled yet sport-specific exercise protocol will elucidate this ergogenic effect. Because IBAs may have different effects on these two groups of athletes, the investigators will measure exercise performance in both female and male elite cyclists. The investigators hypothesize that athletes will perform better during a combination steady-state/sprint exercise task following salbutamol administration.

ELIGIBILITY:
Inclusion Criteria:

* maximal oxygen consumption of ≥60 and ≥55 mL⋅kg-1⋅min-1 or ≥5⋅L⋅min-1 and ≥4⋅L⋅min-1 for men and women

Exclusion Criteria:

* pregnant women
* any history of uncontrolled respiratory or cardiac disease
* smokers
* diabetics

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-01; Primary Completion 2015-11 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Peak Power Output | peak power output of the final 30 seconds of the cycling bout will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Koehle, MD, PhD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Environmental Physiology Laboratory, Vancouver, British Columbia, Canada